CLINICAL TRIAL: NCT06019624
Title: Fresh Takes!: An Evaluation of the Impact of Receiving Fresh Food Boxes on Dietary Intake, Food Insecurity, and Diabetic Control for Individuals With Diabetes or Prediabetes
Brief Title: Fresh Takes!: An Evaluation of the Impact of Receiving Fresh Food Boxes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2023-14791
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes; PreDiabetes; Food Insecurity
Keywords: Diabetes; PreDiabetes; Food Insecurity
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Receipt of Food Box (Active Comparator): Up to 80 individuals with diabetes or prediabetes with a history of food insecurity enrolled in a 6 month program offering free bimonthly fresh food boxes, nutrition education, and individualized support. Each enrolled individual will serve as their own control. The study will evaluate pre and post program changes in reported self-obtained home glucose levels, food security, and dietary intake.
  Interventions: Behavioral: Fresh Takes!
- Cohort 2 Receipt of Food Box (Active Comparator): Up to 80 individuals with diabetes or prediabetes with a history of food insecurity enrolled in a 6 month program offering free bimonthly fresh food boxes, nutrition education, and individualized support. Each enrolled individual will serve as their own control. The study will evaluate pre and post program changes in reported self-obtained home glucose levels, food security, and dietary intake.
  Interventions: Behavioral: Fresh Takes!
- Cohort 3 Receipt of Food Box (Active Comparator): Up to 80 individuals with diabetes or prediabetes with a history of food insecurity enrolled in a 6 month program offering free bimonthly fresh food boxes, nutrition education, and individualized support. Each enrolled individual will serve as their own control. The study will evaluate pre and post program changes in reported self-obtained home glucose levels, food security, and dietary intake.
  Interventions: Behavioral: Fresh Takes!
- Cohort 4 Receipt of Food Box (Active Comparator): Up to 80 individuals with diabetes or prediabetes with a history of food insecurity enrolled in a 6 month program offering free bimonthly fresh food boxes, nutrition education, and individualized support. Each enrolled individual will serve as their own control. The study will evaluate pre and post program changes in reported self-obtained home glucose levels, food security, and dietary intake.
  Interventions: Behavioral: Fresh Takes!

INTERVENTIONS:
Behavioral: Fresh Takes! — Receipt of a fresh produce box, nutritional education and support in a 6 month program

SUMMARY:
Fresh Takes! is a targeted food distribution and nutrition education program offered by Montefiore Bronx Health Collective, a Federally Qualified Health Center located in the South Bronx. The goal of Fresh Takes! is to help reduce food insecurity and prevent progressions to overt diabetes in patients with prediabetes and to help patients with overt diabetes achieve better diabetic control. To that end, participants receive bimonthly fresh food boxes and nutritional support and education over the course of a six-month program.

DETAILED DESCRIPTION:
Diabetes affects approximately one in 10 individuals in the United States and is associated with cardiovascular disease, nerve and retinal damage, and kidney disease. In 2019, it was reported to be the 7th leading cause of death nationally. Unfortunately, diabetes disproportionally affects people of color, those of heavier weight, and those with lower incomes. All of these characteristics are common in residents of the communities served by Montefiore Bronx Health Collective (BHC). Enrolling patients in care at BHC with prediabetes or overt diabetes into Fresh Takes! has the potential to improve short term outcomes and reduce the risk of developing diabetes-associated comorbidities for a highly vulnerable population. The 6-month program has three major components: 1) receipt of a fresh food box twice each month, 2) group nutrition education provided at the time of bimonthly food pickup, and 3) individualized support by a dietician. One of the unique aspects of Fresh Takes! is the provision of a fresh food box to participants. Healthier dietary patterns have been found to be associated with significantly lower risk of developing diabetes and better glycemic control among individuals with diabetes. Yet, little research to date has been conducted on the impact of providing fresh fruits and vegetables on diabetic control for individuals with diabetes or prediabetes.

As an exploratory assessment, following a protocol amendment submitted and approved by the IRB, to determine whether extra education and support is helpful for patients in using all of the contents of the food box, a sub-study was embedded into the existing study by providing an information intervention. As part of this sub-study, all cohort participants will receive individual assessment, education, and a food demonstration and recipe using the contents of the box. Each cohort participant will then be randomized to receive one of the following interventions: 1. Instructions to cut and store vegetables or 2. Instructions to cutting & storing vegetables+ additional recipes customized to the contents of the food box. A block randomization approach to randomize participants to receive the intervention will be used. To avoid contamination, the package will be placed within food delivery packages. This sub-substudy will not impact any of the Outcome Measures in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Be a patient of BHC
* Experienced food insecurity in the previous year

Identified as:

1. having diabetes based on an ICD diagnosis code in the Electronic Medical Record (EMR) or having a less than ideal HbA1c level, defined as >6.4% within the preceding 12 months OR
2. having prediabetes based on an ICD diagnosis code in the EMR or by having a HbA1c level between 5.7% - 6.4% in the preceding 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c levels | From baseline up to 12 months after program completion, up to 18 months total
  Change in HbA1C levels will be evaluated from preintervention to postintervention. Participants' baseline HbA1c values will be abstracted from medical records. The HbA1c value obtained during clinical care closest to the time of enrollment will serve as the baseline value. The HbA1c reading obtained during clinical care closest to the end date of the program will be used as the follow up measure. For participants with prediabetes, blood glucose levels will be measured to see whether HbA1c values have normalized (i.e., HbA1c < 5.7%). Participants with diabetes will be assessed as to whether they have achieved better diabetic control (i.e., reduction of 0.5% from their baseline HbA1c level). Change from baseline group results for prediabetes and diabetes participants within each cohort will be summarized using basic descriptive statistics. Elevated HbA1c levels are a significant risk factor in many disease conditions. Better glycemic control leads to more favorable outcomes.
Change in Food Security | At baseline (intake visit), 3 months, and at 6 months (program completion)
  Change in food security from preintervention to postintervention as measured by the USDA Six-item Short Form of the Food Security Survey. Participant responses are coded as described on the short form and the sum of affirmative responses to the six questions in the module represents the raw score on the scale with a possible scoring range of 0-6 with higher scores being indicative of greater food insecurity. Specifically, an overall score from 0-1 represents high food security; an overall score from 2-4 represents low food security; and an overall score from 5-6 represents very low food security. Group results within each cohort will be summarized.

SECONDARY OUTCOMES:
Change in Fruit and Vegetable Intake | At baseline (intake visit), 3 months, and at 6 months (program completion)
  Change in fruit and vegetable intake form pre- to post-intervention as measured by Fruit and Vegetable module of the Dietary Screener Questionnaire (DSQ-FV). The DSQ-FV consists of 10 questions that queries participants regarding their intake of fruits and vegetables. Responses to the questions are converted to an estimated daily average per participant. Higher fruit and vegetable intake is associated with better glycemic control and better overall health. Change from baseline results for each cohort will be summarized using basic descriptive statistics.
Change in Fruit and Vegetable Consumption | At baseline (intake visit), 3 months, and at 6 months (program completion)
  Change in fruit and vegetable consumption will be objectively assessed using a Veggie Meter®. The Veggie Meter is a validated noninvasive device that uses pressure-mediated reflection spectroscopy (RS) to assess the level of skin carotenoids and provides a comparative output of an individual's skin carotenoid score corresponding to data from the general population. The primary goal is to determine the trajectory of carotenoid responsivity to changes in dietary intake. To avoid measurement error, the multi-measurement mode using an average of 3 measurements of carotenoid score as an in-built part of the device will be used. Participants will insert and retract their finger 3 times and an average score will be determined from the 3 values. Change from baseline results for each cohort will be summarized using basic descriptive statistics. Habitual consumption of fruits and vegetables are correlated with increased Veggie Meter skin carotenoid scores.
Number of Diabetes-related Primary Health Care visits | From baseline up to 12 months after program completion, up to 18 months total
  The number of diabetes-related primary health care visits will be recorded to determine if individuals enrolled in Fresh Takes! have fewer excess visits related to diabetes pre- as compared to post-intervention. Diabetes-related visits will be determined from the electronic medical record (EMR) Diabetes-related visits will be pulled from the Electronic Medical Record (EMR) and defined as visits that have an associated ICD code indicating care for diabetes in the 6 months prior to enrollment. Excess care for this study is defined as having more than one visit for diabetes care in a 6-month period. Group results for each cohort will be summarized.
Change in Emergency Room Utilization | From baseline up to 12 months after program completion, up to 18 months total
  Change in emergency room (ER) utilization will be assessed by the number of emergency room visits to determine if individuals enrolled in Fresh Takes! have fewer emergency room visits related to diabetes pre- as compared to post-intervention. Changes in ER use will be analyzed based on surveys and number of ER visits pulled from the EMR for the 6 months prior to enrollment in Fresh Takes! compared to the number of ER visits for participants in the 6 months following program completion. Change from baseline results for each cohort will be summarized using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hackley, PhD, Study Director — Montefiore Medical Center; Rubayat Qadeer, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Bronx Health Collective, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No data to be shared with other researchers